CLINICAL TRIAL: NCT06977269
Title: Safety and Tolerability of Low Motoneuron Stimulation Via Transcranial Magnetic Stimulation in Spinal Muscular Atrophy
Acronym: STIM-SMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charitable Foundation Children with Spinal Muscular Atrophy (Other)
Collaborators: P.V. Voloshyn Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSMA-INPN-2
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: spinal muscular atrophy; Survival Motor Neuron protein (SMN); Neurofilament (NF); transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TMS arm (Experimental): Stimulation (HF-rTMS) of the primary motor cortex, M1 area of the limbs, at a frequency above 5 Hz and an intensity of 90-100% of the resting motor threshold (RMT), over 10 sessions, up to 2400 stimuli per session.
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation; Diagnostic Test: lumbar puncture

INTERVENTIONS:
Device: High-frequency repetitive transcranial magnetic stimulation — High-frequency repetitive transcranial magnetic stimulation targeting the primary motor cortex (M1) of the limbs, delivered at a frequency above 5 Hz and an intensity of 90-100% of the resting motor threshold, across 10 sessions with up to 2400 stimuli per session, is a standard intervention used in various neurological disorders. However, its effects have not been studied in patients with spinal muscular atrophy (SMA).
  Other Names: HF-rTMS
Diagnostic Test: lumbar puncture — Cerebrospinal fluid sampling to measure SMN protein and neurofilament concentrations before and after the TMS intervention.

SUMMARY:
There is a general physiological rule that any organ or system needs some minimal amount of activity to prevent its atrophy or degeneration. Although the relevance of that rule to exercises in neuromuscular patients and for SMA in particular is not definitely proven, clinical observations seem to support this assumption. Also there are several experimental studies which provide additional support for utility of exercise for SMA.

However, making regular exercises may be very challenging with SMA not only due to physical limitations, but due to psychological either.

While being considered as safe and well tolerated intervention, TMS is able to mimic effects of real physical exercises, at least at the level of low motoneuron, it also provides several advantages. For example, possibility to exercise non-collaborative infants, minimization of psychological motivation impact in adults and/or ability to involve very weak muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of 5q-autosomal recessive SMA confirmed by DNA test.
* Informed consent.
* A minimum score of 1 for Entry Item "A" of the Revised Upper Limb Module (RULM) scale for SMA: "Can use hands to hold pencil or pick up a coin/token or drive a powered chair, use phone key pad"

Exclusion Criteria:

* Subject has severe joint contractures that would affect ability to perform study measures, determined by the study physician.
* Subject has a deconditioned respiratory system, per the discretion of the physician investigator.
* Subject has behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Motor Function Measure Scale | The first assessment will be conducted before the initial TMS session, and the second will be performed one to two days after the final TMS session.
  Motor Function Measure (MFM) scale measurement before and after TMS sessions
Change from Baseline of the Revised Upper Limb Module | The first assessment will be conducted before the initial TMS session, and the second will be performed one to two days after the final TMS session.
  Revised Upper Limb Module (RULM) scale measurement before and after TMS sessions
Change from Baseline of the Hammersmith Functional Motor Scale - Expanded | The first assessment will be conducted before the initial TMS session, and the second will be performed one to two days after the final TMS session.
  Hammersmith Functional Motor Scale - Expanded (HFMSE) measurement before and after TMS sessions
Change from Baseline in the 6-Minute Walk Test | The first assessment will be conducted before the initial TMS session, and the second will be performed one to two days after the final TMS session.
  6-Minute Walk Test (6MWT) measurement before and after TMS sessions

CONTACTS AND LOCATIONS:
Overall Officials: Olena V Pisotska, MD, PhD, Principal Investigator — P.V. Voloshyn Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine; Andriy V Shatillo, MD, PhD, Study Chair — P.V. Voloshyn Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine
Locations (1):
- P.V. Voloshyn Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine, Kharkiv, Kharkivs’ka Oblast’, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR